CLINICAL TRIAL: NCT05636800
Title: Pivotal Study to Assess the Clinical Efficacy and Safety of Microwave Treatment for Actinic Keratosis
Brief Title: Microwave Treatment for Actinic Keratosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blackwell Device Consulting (Industry)
Collaborators: Emblation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMBAK2
Record Dates: First submitted 2022-11-14; First posted 2022-12-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Keratosis, Actinic
Keywords: Actinic Keratosis; Swift System; Microwave; Keratosis; Solar Keratosis; Skin Diseases; Precancerous Conditions; Neoplasms; SCC
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Skin Diseases; Precancerous Conditions; Neoplasms

STUDY DESIGN:
Masking Description: This is an open label study, however, there is a blinded site investigator at each site who will not be aware of the AK lesions that are randomized to treatment. The blinded site investigator will assess resolution and reoccurrence of the AK lesions. Photos of the AK lesions will be taken and these will be reviewed by three independent blinded assessors to assess cosmetic outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Microwave Treatment (Swift System) (Experimental): 3-4 Watts applied locally for up to a 3 second burst to each AK lesion, repeated 3 times per lesion. Burst is defined as a single delivery of microwave energy. There will be approximately 20 seconds between each repeat dose.
  Interventions: Device: Swift System
- No Treatment (No Intervention): No Treatment administered

INTERVENTIONS:
Device: Swift System — Localized microwave energy applied to the distinct AK lesion. Each subject will receive treatment for a maximum of 2 visits (4-week interval between treatment).
  For AK lesions assessed as "Thin" AK (Olsen Grades 1 and 2): Set at 3W and apply locally for up to a 3 second burst and adjust the dose and duration. Repeat on the same AK lesion as is tolerable for the subject (3 repetitions). There will be approximately 20 seconds between each repeat dose.
  For AK lesions assessed as "Thick" AK (Olsen Grade 3): Set at 4W and apply locally for up to a 3 second burst and adjust the dose and duration. Repeat on the same AK lesion as is tolerable for the subject (3 repetitions).
  As the AK lesions may be larger than 3mm in diameter, the dose administered to one AK lesion may require overlapping applications with the applicator tip. Ensure there is approximately 20 seconds between each repeat dose administered
  Arms: Microwave Treatment (Swift System)

SUMMARY:
This is a randomized, controlled, multi-center trial in subjects diagnosed with Actinic Keratosis (AK) where each subject serves as their own control. The trial will be conducted at 2 sites, one in Germany and one in the United States. Approximately 60 subjects will be randomized to ensure 51 subjects complete the study.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the efficacy of the Swift Microwave Treatment on resolution of Actinic Keratosis lesions.

The secondary objectives of this trial is to evaluate the efficacy, safety and tolerability of Swift Microwave treatment as a therapy for Actinic Keratosis (AK).

Eligible subjects who provide written informed consent and have 10, 12 or 14 distinct Actinic Keratosis lesions located on their scalp or hands will be randomized onto the study. Randomization of AK lesions will be stratified by side. Subjects will be randomized to treatment on half the number of AK lesions mapped located on their scalp or hands. The mapped AK lesions not randomized for treatment will receive no treatment (control).

The microwave energy applied by the Swift device will be applied to the randomized AK lesion sites for up to 2 treatments, spaced out by a 4-week interval. Follow-up is 2-months after the first treatment is administered where the AK lesions are assessed for resolution. Further follow-up visits occur at 4-months, 6-months and 12-months after the first treatment was administered where the AK lesions will be assessed for resolution or reoccurence.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age 18-85 years inclusive (EU); 22-85 years inclusive (US).
4. AK lesions for randomization in this study: Clinical diagnosis by a dermatologist of precancerous Actinic Keratosis.
5. Cutaneous location.
6. 10, 12 or 14 distinct AK lesions (3-6mm in diameter inclusive), for randomization in this study, located on the subjects' scalp or hands (AK lesions on the scalp and hands for randomization cannot be mixed).

   * There must be at least 2 AK lesions on the left and right side of the scalp or left and right hand.
   * An even number of distinct AK lesions (10, 12 or 14) are to be selected.
   * The maximum possible number of available distinct AK lesions should be selected (10, 12 or 14).
   * The subject may present with any number of AK lesions, however only 10, 12 or 14 distinct AK lesions will be selected for randomization. For example, if a subject presents with 21 AK lesions, an even number of distinct AK lesions are to be selected (i.e. 14 distinct AK lesions with at least 2 distinct AK lesions on the left and right side of the scalp or left and right hand).
7. If currently receiving treatment for Actinic Keratosis, agree to stop their current medication for at least 28 days prior to the start of study treatment.
8. Agrees to refrain from using any other Actinic Keratosis products or treatments during the study period, unless specified by the Investigator.
9. Agrees to refrain from using any topical metallic or ionic treatment (e.g., aluminum chloride, silver nitrate, zinc oxide) during the study period.
10. Free of any disease state or condition which, in the investigator's opinion, could impair evaluation of AK or could expose the subject to an unacceptable risk by study participation.
11. Able to perform study assessments.

Exclusion Criteria:

1. AK lesions at potential treatment sites on lip, nose crease, near eyes or ear.
2. Confluent AK associated with field change at potential treatment sites.
3. Fewer than 2 AK lesions on the left and right side of the scalp or left and right hand.
4. AK lesions at potential treatment sites assessed as clinically ambiguous.
5. Implantable Cardioverter Defibrillator (ICD), pacemaker or other implantable electronic devices.
6. Metal implants at site of treatment.
7. Known allergy or intolerance to microwave therapy.
8. Unstable co-morbidities (cardiovascular disease, active malignancy, vasculopathy, inflammatory arthritis).
9. Previous history of skin cancer in the study treatment or observation area.
10. Previous history of squamous cell carcinoma (SCC) or keratoacanthoma (KA) in any location.
11. Pregnancy or breast feeding.
12. Participating in another interventional study or have done so within the last 30 days.
13. Anticipated relocation or extensive travel outside of the local study area preventing compliance with study procedures.
14. Circulatory conditions affecting the acral areas - peripheral vascular disease, peripheral ischemia, vasculitis, Raynaud's, or related conditions.
15. Peripheral neuropathy.
16. Subject who is immunosuppressed (organ transplant recipients, hematologic malignancies, HIV).
17. Subject who has had any topical metallic or ionic treatment (e.g, aluminum chloride, silver nitrate, zinc oxide) within the last 6 months at potential treatment sites.
18. Subjects with AK on the scalp and who have hearing aid(s) and are unable or unwilling to remove hearing aids prior to microwave treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with treatment success of Actinic Keratosis at 2 months following Swift Microwave treatment. | 2 months post first treatment
  Definition:
  Treatment Success: complete clearance of ≥75% Actinic Keratosis lesions treated per subject, i.e., at least 75% of the AK lesions treated are fully cleared (not partially cleared).

SECONDARY OUTCOMES:
Proportion of subjects with treatment success of Actinic Keratosis following Swift Microwave treatment. | 4 and 6 months post first treatment
Proportion of subjects with 100% clearance of Actinic Keratosis following Swift Microwave treatment | 2, 4 and 6 months post first treatment
Percentage of Actinic Keratosis lesions cleared across all study lesions following Swift Microwave treatment | 2, 4 and 6 months post first treatment
OCT Analysis as assessed by an AK Classification System | Baseline and 2, 4 and 6 months post first treatment
  AK Lesions classified as Not Present, AK I (Grade I mild), AK II (Grade II, moderate) or AK III (Grade III severe)
Proportion of subjects with reoccurrence of any Actinic Keratosis lesions at 6 months, as classified by the blinded site investigator. The subject's AK lesion must be classified as completely resolved at 2 months to be considered a reoccurrence. | 6 months post first treatment
Level of pain during treatment using a severity scale | Treatment 1 (Day 0), Treatment 2 (Day 28)
  The subject is asked to rate the worst pain experienced during treatment as None, Mild, Moderate or Severe
Level of pain after treatment using a severity scale | Treatment 1 (Day 0), Treatment 2 (Day 28)
  The subject is asked to rate the worst pain experienced during the 10 minute period after treatment is completed as None, Mild, Moderate or Severe
Duration of pain after treatment using a time period scale | Treatment 1 (Day 0), Treatment 2 (Day 28)
  For subjects who experienced pain after treatment, the subject is asked to rate the duration of pain experienced during the 10 minute period after treatment using the following time period scales: a few seconds, up to 1 minute, up to 2 minutes, up to 3 minutes, Still Sore.
Difference in cosmetic outcomes between treated and non-treated Actinic Keratosis as classified by the independent blinded assessors using a grading system | 2, 4 and 6 months post first treatment
  Photographs of each treated and non-treated AK lesion will be assessed by the independent blinded assessors for cosmetic outcome as "excellent" (slight redness or pigmentation change), "good" (moderate redness or pigmentation change), "fair" (slight-to-moderate scarring, atrophy or induration), or "poor" (extensive scarring, atrophy or induration). Each assessment compares the photos taken at the current visit against the photos taken at the previous visit. The assessments by each independent blinded assessor is recorded separately.
Severity and occurrence of Adverse Events | Up to 12 months post first treatment
Evaluation of Patient Reported Outcome (PRO) at baseline and 6 months post first treatment using a rating scale | Baseline and 6 months post first treatment
  At Baseline, the subject will be asked to rate how their AK lesions affect their daily activities, lifestyle and mood as: none, mild, moderate and severe.
  At 6-months post first treatment, the subject will be asked to rate how their daily activities, lifestyle and mood are now affected, when compared to before study treatment as: significantly better, better, unchanged, worse, significantly worse.
  The results at baseline and at 6 months post first treatment will be evaluated.
Evaluation of Quality of Life (QoL) questionnaires at baseline and 6 months post first treatment using the Dermatology Life Quality Index (DLQI) questionnaire | Baseline and 6 months post first treatment
  The DLQI questionnaire measures how the AK lesions have affected the subject's life over the past week. The score at baseline and at 6 months post first treatment will be evaluated.
Evaluation of Cosmetic Outcome at 6 months post first treatment using a rating scale | 6 months post first treatment
  The subject will be asked to rate the AK lesions that were treated compared to before treatment as: significantly better, better, unchanged, worse, significantly worse.
Long term follow-up of subjects with reoccurrence at 12 months as classified by the blinded site investigator | 12 months post first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dirschka, Principal Investigator — CentroDerm GmbH, Heinz-Fangman-Strasse 57, 42287 Wuppertal (Barmen), Germany; Dr Waibel, Principal Investigator — Miami Dermatology and Laser Institute, Miami, Florida, United States, 33173
Locations (2):
- Miami Dermatology and Laser Institute, Miami, Florida, United States
- Centroderm GmbH, Wuppertal, Germany